CLINICAL TRIAL: NCT02781987
Title: Changhai Hospital, the Second Military Medical University
Brief Title: Incidence and Risk Factor of Post-ERCP Pancreatitis in Chronic Pancreatitis
Status: Completed | Type: Observational
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhuan Liao, associate professor, Changhai Hospital
Other Study IDs: PEP-CP; 81470884 (Other Grant/Funding Number: National Natural Science Foundation of China); 81422010 (Other Grant/Funding Number: National Natural Science Foundation of China); 81270541 (Other Grant/Funding Number: National Natural Science Foundation of China); 13QA1404600 (Other Grant/Funding Number: the Shanghai Rising-Star Program)
Record Dates: First submitted 2016-05-18; First posted 2016-05-25 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Post-ERCP Acute Pancreatitis

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- CP group: Those patients with chronic pancreatitis underwent ERCP for pancreatic stone clearance, pancreatic stent placement, etc..
  Interventions: Other: chronic pancreatitis
- BD group: Those patients with biliary ductal disease, such as choledocholithiasis, underwent ERCP to relieve outflow obstruction of the common bile duct.

INTERVENTIONS:
Other: chronic pancreatitis — patients with chronic pancreatitis
  Groups: CP group

SUMMARY:
The purpose of this study is to compare the incidence of post-ERCP pancreatitis (PEP) in chronic pancreatitis (CP) patients to that in biliary disease patients, to determine whether CP patients in early clinical stage have a higher PEP incidence, and to identify the predictive and protective factors for PEP in chronic pancreatitis patients.

DETAILED DESCRIPTION:
Analysis of patients with chronic pancreatitis (CP group) and biliary disease (BD group) in Changhai Hospital from January 2011 to May 2015 were conducted. Difference of PEP incidences between BD group and CP group, as well as between M-ANNHEIM subcategories were calculated by chi-square test or Fisher's exact test. The predictive and protective factors for PEP were investigated by univariate and multivariate analysis.

ELIGIBILITY:
Inclusion Criteria:

* patients with an endoscope inserted to cannulate the pancreatic/biliary duct were included.

Exclusion Criteria:

* patients in whom the papilla of Vater was not reached;
* patients who underwent stent removal procedures without ductal cannulation;
* patients in whom the intubation was failed.

Ages: 5 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Chronic pancreatitis patients underwent ERCP from January 2011 to May 2015 in Changhai Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 2028 (Actual)
Dates: Start 2011-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Numbers of chronic pancreatitis patients with post-ERCP pancreatitis, diabetes mellitus, steatorrhea, previous pancreatitis, previous PEP, pancreatic divisum, jaundice, ESWL, pancreatic duct stone, drainage and minor papilla pancreatogram. | 8 months

SECONDARY OUTCOMES:
Numbers of biliary disease patients with post-ERCP pancreatitis, previous pancreatitis and previous PEP. | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Zhao-shen Li, Study Chair — Changhai Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zhao ZH, Hu LH, Ren HB, Zhao AJ, Qian YY, Sun XT, Su S, Zhu SG, Yu J, Zou WB, Guo XR, Wang L, Li ZS, Liao Z. Incidence and risk factors for post-ERCP pancreatitis in chronic pancreatitis. Gastrointest Endosc. 2017 Sep;86(3):519-524.e1. doi: 10.1016/j.gie.2016.12.020. Epub 2017 Jan 4. PMID 28062312